CLINICAL TRIAL: NCT06017492
Title: Effects of Video-assisted Discharge Education of Day Surgery Patients on the Perception of Quality of Discharge Teaching and Satisfaction With Nursing Care
Brief Title: Effects of Video Use on Quality of Discharge Teaching and Patient Satisfaction in Day Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Sandra Chirota Akire, Principal Investigator, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PE in day surgery patients
Record Dates: First submitted 2023-08-14; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Patient Satisfaction; Quality of Care
Keywords: Day care surgery; Patient education; Discharge teaching; video-assisted patient education; Ambulatory surgery; Nursing care
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized in a one- to-one intervention allocation to the intervention (n = 86) or usual hospital method (n=86) group at the time of consent.
Who Masked: Participant
Masking Description: Allocation concealment will be blinded and performed in the order of recruitment using a computerized generated allocation method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital Patient Education Method (No Intervention): Control Group:
  Implementation will be carried out in 2 phases; Phase 1(intervention): participants will receive hospital-based patient education method(printouts, verbal instruction). This intervention will be carried out in a 2 weeks period; starting 2 weeks before day surgery and ending after day surgery has been carried out.
  Phase 2 (post test): In this part, participants will be asked to answer questions in the in the descriptive data, the Quality of Discharge Teaching Scale (QDTS) and Patient Satisfaction with Nursing Care Quality Questionnaire (PSNCQQ). The questionnaire will be printed and distributed to participants after Day Surgery. The questionnaire will also be in Google form format and sent to emails of participants who are not physically present at the clinic.
- Audio-Visual Patient Education Method (Experimental): Implementation will be carried out in 2 phases; Phase 1(intervention): participants will recieve video assisted teaching as patient education method. Series of short videos will be played for the participants to watch and also sent to their phones through Whatsapp application or email. This intervention will be carried out in a 2 weeks period; starting 2 weeks before day Surgery and ending after day Surgery has been carried out.
  Phase 2(post test): In this part, participants will be asked to answer questions in the in the descriptive data, the Quality of Discharge Teaching Scale (QDTS) and Patient Satisfaction with Nursing Care Quality Questionnaire (PSNCQQ). The questionnaire will be printed and distributed to participants after Day Surgery. The questionnaire will also be in Google form format and sent to emails of participants who are not physically present at the clinic.
  Interventions: Behavioral: video assisted discharge teaching

INTERVENTIONS:
Behavioral: video assisted discharge teaching — Patients will be educated using the video assisted discharge teaching. The educational content will be in English and will focus on the following topics: surgical process, medication use complication after surgery, pain management, wound care, nutrition, self-care after, surgery, home care after surgery and situations to refer to a physician.
  Arms: Audio-Visual Patient Education Method

SUMMARY:
this study is aimed to determine the effects of video-assisted discharge education of day surgery patients on the perception of quality of discharge Study Hypothesis include the following; H1: The day surgery patients who were exposed to the video-assisted discharge educational intervention will have higher perception on quality of discharge teaching, compared with those who were not exposed to the educational intervention.

H2: The day surgery patients who were exposed to the video-assisted discharge educational intervention will have enhanced satisfaction with nursing care quality, compared with those who were not exposed to the educational intervention

DETAILED DESCRIPTION:
The goal of patient education in Daycare surgery is to improve overall patient outcome and satisfaction. Comprehensive patient assessment, putting into consideration patient's needs and expected postoperative difficulties, will help nurses in understanding types of patient education strategies that can be used in order to promote better individualized quality discharge education which in turn leads to the best postoperative outcomes (Quemby& Stocker, 2014; Jaensson, Dahlberg & Nilsson, 2019).

Although there are various studies showing the effects of video assisted patient education, there are only a few clinical studies concentrating on Day care Surgery patients and none in Turkey. Therefore, we will examine the effect of video-assisted teaching in relation to discharge planning, quality of nursing care and overall patient satisfaction in Day Care Surgery patients' group. The result of this study may guide for development of the educational strategies for Day Care Surgery patients.

The study will be conducted in Jinepol Women's Health and IVF clinic in Turkey Jinepol.

The study aims to recruit one hundred and seventy two (172) patients into the program. 86 participants will be selected in each group, using the simple random sampling method from December 2022- December 2023

Study tools:

A descriptive data form, The Quality of Discharge Teaching Scale (QDTS) and Patient Satisfaction with Nursing Care Quality Questionnaire (PSNCQQ) will be used in data collection. The descriptive data form which will provide information about patients' gender, nationality, age, type of surgery, educational level and occupation will be made by the researcher. Ethical approval was obtained from Institutional Reviews Board (IRB) of Near East University Hospital. In addition, informed consent from the patients and organizational permission will be obtained. An institutional permission was obtained from the management of Jinepol Women's Health and IVF Clinic. Since Permission has already been granted by the authors of the Quality of Discharge Teaching Scale and the Patient Satisfaction with Nursing Care Quality Questionnaire (PSNCQQ) to use the scales, no further permission will be required.

Statistical Package of SocialSciences (SPSS) software version 20.0 will be used to analyze the collected data. Descriptive statistics (ie, means, standard deviations, and frequencies and percentages) will be used to calculate for all patient characteristics and response items. A chi-square test and independent T test will be used to determine the hypothesis either null or alternate at a significant level of p < 0.05.

Evaluation of The Quality of Discharge Teaching Scale (QDTS) are as follows; 10: Excellent

8 and 9 = very good

6 and 7 = good

5 = neutral

3 and 4 = fair

1 and 2 = poor

0 = none/not at all

The Mean of content and delivery subscales scores will be calculated separately.

Evaluation of the Patient Satisfaction with Nursing Care Quality Questionnaire (PSNCQQ) are as follow; 5 = Excellent

4 = very good

3 = good

2 = fair

1 = poor.

The Mean and Standard deviation of items will be calculated

ELIGIBILITY:
Inclusion Criteria:

* Female patients, who understand English, have had day care surgery.

Exclusion Criteria:

* Patients less than 18 years of age
* Patients who do not understand or cannot read in English
* Patients with complications
* Patients who undergo surgery for oncological reasons
* Patients whose hospital stay was longer than 24 hours.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Effects of discharge education of day surgery patients on the perception of quality of discharge | up to 2 days after day surgery procedure
  effects of video assisted discharge education of day surgery patients on the perception of quality of discharge teaching as measured using the Quality of Discharge Teaching Scale (QDTS) by Marianne Weiss (weiss, 2022). the scale measures perception of patients' quality of discharge teaching which has been provided by nurses during the preparation for discharge. it is a 0 - 10 scale (0 = none, 10= Excellent), with higher scores reflecting a greater amount of information recieved and higher quality of discharge teaching
Effects of discharge education of day surgery patients on Satisfaction with Nursing Care | up to 2 days after day surgery procedure
  The Patient Satisfaction with Nursing Care Quality Questionnaire 2005 (PSNCQQ) will be used to assess satisfaction of nursing care after day surgery. A 5- point Likert scale ranging from 'excellent' (5) to 'poor' (1) is used in each item of the Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra C Akire, PhD, Principal Investigator — Near East University
Locations (1):
- Jinepol Women's Health and IVF Clinic, Levent, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No